CLINICAL TRIAL: NCT01605773
Title: Repaglinide Versus Glyburide: Comparitive Effect on Postprandial Lipemia: An Open-labeled, Randomized, Parallel Group Study in Patients With Type 2 Diabetes
Brief Title: Effect of Repaglinide on Postprandial Lipemia in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-2137
Record Dates: First submitted 2012-05-16; First posted 2012-05-25 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- repaglinide (Experimental)
  Interventions: Drug: repaglinide
- glyburide (Active Comparator)
  Interventions: Drug: glyburide

INTERVENTIONS:
Drug: repaglinide — Dose individually adjusted and conducted according to labeling
  Arms: repaglinide
Drug: glyburide — Dose individually adjusted and conducted according to labeling
  Arms: glyburide

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to compare the effect of repaglinide on postprandial lipemia in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with type 2 diabetes currently treated with diet and exercise alone (HbA1c below 10%)
* Subjects with type 2 diabetes treated with sulphonylurea (HbA1c below 8.5%)
* Males or non-pregnant, non-lactating females
* Subjects should have normal renal function

Exclusion Criteria:

* Type 1 or other specific causes of diabetes
* Marked symptomatic diabetes
* Uncontrolled treated/untreated hypertension
* Known or suspected allergy to the trial products or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2001-11-08; Primary Completion 2003-03-13 (Actual); Study Completion 2003-03-13 (Actual)

PRIMARY OUTCOMES:
Triglyceride levels post standardised fat tolerance test

SECONDARY OUTCOMES:
Incidence of hypoglycemic episodes
Change in HbA1c (glycosylated haemoglobin A1c)
Change in FPG (fasting plasma glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Houston, Texas, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com